CLINICAL TRIAL: NCT00708266
Title: A Mono-Centre Randomized Study to Investigate the Effect of Elevated Plasma Fatty Acid Concentrations on Cytokines in Interstitial Fluid of Subcutaneous Adipose Tissue
Brief Title: The Influence of Fatty-Acids on Systemic and Subcutaneous Cytokines
Acronym: TNF4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Thomas R. Pieber, Medical University Graz
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: TNF4
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-06

CONDITIONS: Obesity; Type 2 Diabetes Mellitus
Keywords: Obesity; Diabetes; Non-esterified fatty acids; Cytokines; Inflammation; Subcutaneous fat; Adipose tissue
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Diabetes Mellitus; Inflammation | interventions — safflower oil, soybean oil, lecithin emulsion; Saline Solution; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- V2 (Placebo Comparator): 28 hours continuous saline venous infusion.
  Interventions: Device: Openflow microperfusion catheter; Other: 0.9% Saline Solution
- V3 (Experimental): 28 hours continuous lipid-heparin venous infusion.
  Interventions: Device: Openflow microperfusion catheter; Dietary Supplement: Intralipid 20%

INTERVENTIONS:
Device: Openflow microperfusion catheter — Macro-perforated, double lumen catheter used to withdraw interstitial fluid samples from different tissues.
  Other Names: No other names registered.
Dietary Supplement: Intralipid 20% — Lipid emulsion used in clinical practice as supplementary intravenous nutrition. 28 hours venous infusion during the "treatment" study visits.
  Other Names: Liposyn
  Arms: V3
Other: 0.9% Saline Solution — 0.9% sodium chloride solution, used in clinical practice for venous hydration. 28 hours infusion during the "control" study visits.
  Other Names: - Saline; - 0.9% Sodium Chloride
  Arms: V2

SUMMARY:
This is a mono-center randomized controlled trial to be performed in the Center of Medical Research (ZMF) at Medical University Graz and is composed by one screening visit (V1) and two study visits (V2 and V3). In the visit V1, complete medical examination will be performed and blood samples will be withdrawn to check overall conditions of the healthy volunteers. Those who accomplish the necessary conditions will be enrolled in the trial to receive either saline or lipid-heparin solutions in a randomized, cross-over design during visits V2 and V3. Volunteers will arrive at ZMF after overnight fasting, when two venous catheters will be placed in forearm veins. One venous catheter will be used for continuous infusion of lipid-heparin solution (Intralipid 20%, 40 ml/h, Fresenius Kabi plus Heparin 250U/h, IMMUNO Baxter AG) or saline, and Inulin (Inutest 25%, Fresenius Kabi). The second venous catheter will be used for blood sampling (arterialized venous blood). Subsequently, two open flow microperfusion (OFM) macro-perforated catheters will be inserted in the subcutaneous tissue of abdominal wall for continuous sampling of interstitial fluid. Study visits will last for 28 hours for continuous sampling, with four additional hours for observation after infusion discontinuation, during visits V2 and V3. Concentrations of different cytokines, non-esterified fatty-acids, insulin, glucose, triglycerides and inulin will be retrospectively quantified in the frozen samples.

The primary hypothesis is that cytokine concentrations in subcutaneous tissue and/or in circulation can be modified by lipid-heparin infusion.

DETAILED DESCRIPTION:
1. General

   Subjects will be selected to participate in the protocol during study visit 1 according to the inclusion and exclusion criteria. Subsequently they will be randomly assigned to receive continuously an intravenous infusion of 0.9% saline or a lipid-heparin solution (Intralipid 20%, 40 ml/h, Fresenius Kabi plus Heparin 250U/h, IMMUNO Baxter AG) during 28 hours at study visits V2 and V3. For the study visit 3, subjects who first received 0.9% saline in the previous visit, will receive intravenously Intralipid 20% and vice versa.
2. Visit Procedures

   2.1. Screening Day (Visit 1)

   Volunteers will receive overall information about the study and sign in the written informed consent. Every subject will receive an assignment number according to the inclusion sequence. Physical examination and blood withdrawal shall be performed and data will be recorded in the Case Report Form (CRF) as follows:
   * Inclusion/exclusion criteria
   * Demographic data, medical history and concomitant medication
   * Physical examination
   * Vital signs
   * Body weight and height, Body mass index (BMI), waist and hip circumference and waist-to-hip ratio
   * Blood blood count, hematocrit, hemoglobin, C-reactive protein, free fatty acids, cholesterol, triglycerides, sodium, potassium, calcium
   * Pregnancy test for female subjects of childbearing potential.

   2.2. Study day (Visit 2 and 3)

   During each study visit subjects shall arrive at 7:00 AM at ZMF (Center of Medical Research, Medical University Graz) after an overnight fasting period of 12 hours. A pregnancy test for female subjects of childbearing potential will be performed in the morning of each study day. Two short polyethylene catheters will be inserted in antecubital veins of both arms. A first venous cannula will be exclusively used for blood sampling and the arm will be placed in a thermo regulated box (Hot-Box) to be maintained warmed at a temperature of 50°C over the whole study period. The second venous cannula will be used for infusion of saline or lipid-heparin solution and inulin.

   At 8:00 AM, the infusion of saline or Intralipid solution will be started. At the same time point a continuous infusion of inulin via syringe infusion pump will be started with a 50mg/Kg bolus and maintained at a continuous rate of 0.250 x Creatinin Clearance mg/min, until the end of the study period.

   At 11:00 AM, OFM catheters will be inserted in the periumbilical area of each subject. To prevent important delays in sampling from subcutaneous tissue, the afferent loop for the catheter will be previously filled with the perfusate solution. Eight milliliters of a sterile isotonic solution (ELO MEL isoton, Fresenius Kabi, Austria) commonly used as intravenous infusion added with 2.0ml autologous serum previously withdrawn from each volunteer and prepared under straight sterile conditions will be used as the perfusate solution for the OFM catheters. Peristaltic pumps will start to run at 12:00 AM to infuse the perfusate solutions at a perfusion rate (push-pull mode) of 1µl/min until 12:00 AM in the following day. Effluent samples from subcutaneous tissue will be collected at regular time-intervals and venous blood sampling will be performed in parallel.

   The subjects will be maintained under fasting conditions during the whole study period. They shall stay in the research center facilities for a four-hours observation period after the study procedures have finished. At this time they will receive a complete meal and additional blood samples will be withdrawn to access blood glucose and aPTT (activated partial tromboplastin time). Normal values have to be ensured before the volunteers are allowed to leave.
3. Measurements

3.1. Cytokines

Cytokine concentrations will be measured in effluent and serum samples using a multiplexed flow cytometric bead-based ELISA assay (LUMINEX®100s System, Luminex Corporation, Texas, USA). The following substrates will be accessed by this method:

* C-reactive protein
* Interleukin 6 (IL-6)
* Interleukin 10 (IL-10)
* CCL2/MCP-1
* Serpin E1/PAI-1
* Tumor Necrosis Factor alpha (TNF-alpha)
* Adiponectin

3.2. Insulin

Insulin concentrations in effluent and plasma samples will be measured by Joanneum Research Laboratory using solid-phase two-site ELISA (Mercodia, Uppsala, Sweden).

3.3. Inulin

Inulin will be measured by Joanneum Research Laboratory, using a fully enzymatic method.

3.4. Glucose

Glucose concentration in arterialized blood samples will be measured in duplicate using two Beckman Glucose Analyzer 2 (Beckman Instruments Inc., Fullerton, CA).

3.5. Non-esterified fatty acids (NEFA)

NEFA concentrations will be measured in plasma using a colorimetric and enzymatic method.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed before any study activities.
* Age of 18 years old or above.
* A body mass index (BMI) within the limits of 18.5 to 24.9 (normal range).

Exclusion Criteria:

* Any clinical signs of acute or chronic inflammation detectable during study visit 1.
* Severe acute or chronic diseases (e.g. acute respiratory tract infection, systemic lupus erythematosus, rheumatoid arthritis).
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
* Use of any vasoactive substances (e.g. anti-hypertensive drugs), immune-suppressant or anti-inflammatory drugs (e.g. corticosteroids, aspirin, other COX2 inhibitors) or anti-coagulation treatment.
* Diseases of the skin which could interfere with catheter insertion in the abdominal wall.
* Pregnancy in women subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Concentrations of IL-6 measured in effluent samples from subcutaneous tissue. | 24 hours of interstitial fluid sampling

SECONDARY OUTCOMES:
Concentrations of all other cytokines measured in effluent samples from subcutaneous tissue. | 24 hours of interstitial fluid sampling.
Cytokine concentrations measured in serum samples. | 24 hours sampling during the experiment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Pieber, M.D., Principal Investigator — Medical University Graz, Graz, Austria
Locations (1):
- Medical University Graz - Clinical Research Center, Graz, Styria, Austria